CLINICAL TRIAL: NCT01514500
Title: First Human Dose Trial of NNC0195-0092 (Somapacitan) in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: NN8640-3915; U1111-1119-0539 (Other: WHO); 2011-000146-38 (EudraCT Number)
Record Dates: First submitted 2012-01-13; First posted 2012-01-23 (Estimated); Last update posted 2020-12-24 (Actual); Status verified 2020-12

CONDITIONS: Growth Hormone Disorder; Adult Growth Hormone Deficiency; Growth Hormone Deficiency in Children; Healthy
MeSH Terms: conditions — Dwarfism, Pituitary | interventions — somapacitan; NNC0195-0092

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Single dose (SD) (Experimental): Single dose administered s.c. (subcutaneously, under the skin). Escalation to the next dose level will be based on safety evaluation
  Interventions: Drug: somapacitan; Drug: placebo (somapacitan)
- Multiple dose (MD) (Experimental): Multiple doses administered s.c. (subcutaneously, under the skin). All subjects will be dosed four times with a dosing frequency of once weekly. Escalation to the next dose level will be based on safety evaluation
  Interventions: Drug: somapacitan; Drug: placebo (somapacitan)

INTERVENTIONS:
Drug: somapacitan — Administered s.c. (subcutaneously, under the skin)
  Other Names: NNC0195-0092
Drug: placebo (somapacitan) — Single or multiple placebo doses administered s.c. (subcutaneously, under the skin)

SUMMARY:
This trial is conducted in Europe. The aim of this trial is to assess safety, tolerability, pharmacokinetics (the exposure of the trial drug in the body) and pharmacodynamics (the effect of the investigated drug on the body) of NNC0195-0092 (somapacitan) compared to placebo in healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, non-smoking male subjects
* BMI (body mass index) between 18.0 and 28.0 kg/m^2, both incl.
* Body weight 50 to 100 kg, both incl.

Exclusion Criteria:

* Strenuous exercise within 4 days prior to dosing
* Receipt of any investigational medicinal product within 3 months prior to randomisation

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 105 (Actual)
Dates: Start 2012-01-16 (Actual); Primary Completion 2013-03-18 (Actual); Study Completion 2013-03-18 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events (Single Dose) | From first administration of trial product and up until day 40
Incidence of adverse events (Multiple Dose) | From first administration of trial product and up until day 49

SECONDARY OUTCOMES:
Area under the NNC0195-0092 (somapacitan) serum concentration-time curve | From 0 to 168 hours
Area under the NNC0195-0092 (somapacitan) serum concentration-time curve (SD part only) | From 0-240 hours
Area under the NNC0195-0092 (somapacitan) serum concentration-time curve (SD part only) | up to day 40
Maximum serum concentration (Cmax) for NNC0195-0092 (somapacitan) | up to day 40
Area under the IGF-I (insulin-like growth factor-I) serum concentration-time curve | From 0-168 hours
Area under the IGF-I (insulin-like growth factor-I) serum concentration-time curve (SD part only) | From 0-240 hours
Maximum serum concentration (Cmax) for IGF-I | up to day 40
Area under the IGFBP-3 (insulin-like growth factor binding protein-3) serum concentration-time curve | From 0-168 hours
Area under the IGFBP-3 (insulin-like growth factor binding protein-3) serum concentration-time curve (SD part only) | From 0-240 hours
Maximum serum concentration (Cmax) for IGFBP-3 | up to day 40
Number of injection site reactions | From first administration of trial product and up until day 40 (SD part)
Number of injection site reactions | From first administration of trial product and up until day 49 (MD part)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR,1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Neuss, Germany

REFERENCES:
- [Background] Juul Kildemoes R, Hojby Rasmussen M, Agerso H, Overgaard RV. Optimal Monitoring of Weekly IGF-I Levels During Growth Hormone Therapy With Once-Weekly Somapacitan. J Clin Endocrinol Metab. 2021 Jan 23;106(2):567-576. doi: 10.1210/clinem/dgaa775. PMID 33313798
- [Derived] Juul RV, Rasmussen MH, Agerso H, Overgaard RV. Pharmacokinetics and Pharmacodynamics of Once-Weekly Somapacitan in Children and Adults: Supporting Dosing Rationales with a Model-Based Analysis of Three Phase I Trials. Clin Pharmacokinet. 2019 Jan;58(1):63-75. doi: 10.1007/s40262-018-0662-5. PMID 29671202
- [Derived] Rasmussen MH, Olsen MW, Alifrangis L, Klim S, Suntum M. A reversible albumin-binding growth hormone derivative is well tolerated and possesses a potential once-weekly treatment profile. J Clin Endocrinol Metab. 2014 Oct;99(10):E1819-29. doi: 10.1210/jc.2014-1702. Epub 2014 Jul 11. PMID 25013997
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com